CLINICAL TRIAL: NCT01631526
Title: Open Clinical Trial to Validate a Short-term Vitamin D Loading and Maintenance Dose Protocol in People With Advanced Lung Cancer
Brief Title: Vitamin D Loading Dose in Advanced Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, John Hoffer, Professor of Medicine, McGill University, Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC12-053
Record Dates: First submitted 2012-06-27; First posted 2012-06-29 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Lung Cancer
Keywords: Lung cancer; vitamin D; pharmacokinetics
MeSH Terms: conditions — Lung Neoplasms | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin D (Experimental): vitamin D 20,000 IU per day for 2 weeks followed by 10,000 IU per day for a further 7 days
  Interventions: Dietary Supplement: vitamin D

INTERVENTIONS:
Dietary Supplement: vitamin D — vitamin D3 20,000 IU per day for 14 days followed by 10,000 IU per day for a further 7 days

SUMMARY:
Hypovitaminosis D is highly prevalent in people with lung cancer, and may have adverse clinical consequences. The long and variable pharmacokinetic half-life of vitamin D makes prompt vitamin D replacement problematic. This is an open, one-armed therapeutic intervention using a loading dose of vitamin D that will be predicted to increase plasma 25-hydroxyvitamin D concentrations of every patient well into the normal range (> 100 nmol/L) within 2 or 3 weeks and monitored after 2 and 3 weeks of loading and maintenance dose. Preliminary data will also be obtained to identify potentially clinical important outcome benefits for future investigation. The outcomes are

1. plasma 25OHD concentration
2. Vitamin D binding protein and other plasma concentrations
3. Mood and symptom

ELIGIBILITY:
Inclusion Criteria:

1. Any patient with advanced lung cancer whether or not receiving specific anti-cancer therapy
2. Mentally competent (but need not be fluent in French or English if capable neutral translator available)
3. Self report of reduced food intake and/or involuntary weight loss of any extent at time of enrollment: does not have to be documented

Exclusion Criteria:

1. Current diagnosis of primary hyperparathyroidism
2. Nephrocalcinosis
3. Current or suspected active tuberculosis, histoplasmosis, sarcoidosis, or other granulomatous disease
4. Current using a vitamin D supplement providing > 1000 IU/day
5. Current prescribed calcitriol in any dose
6. History of extensive sunlight exposure (> 30 min summer sunlight exposure per day for more than 5 days per week) in previous 3 months
7. Expected to die within next 2 months
8. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-06; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Plasma 25-hydroxyvitamin D concentration | 3 weeks
  Plasma 25OHD concentration measured within 24 h prior to commencing vitamin D therapy, and again after 14 and 21 days of continuous vitamin D therapy

SECONDARY OUTCOMES:
Mood | 3 weeks
  Two validated brief mood assessment questionnaires measured
  1. On two occasions (one week apart) at baseline prior to staring therapy
  2. After 2 weeks of therapy
  3. After 3 weeks of therapy
Symptoms | 3 weeks
  As with mood questionnaire, a symptom questionnaire (Edmonton Symptom Assessment System) will be administered two times (one week apart) prior to starting vitamin therapy and after 14 and 21 days of continuous vitamin D administration

CONTACTS AND LOCATIONS:
Locations (1):
- Brojde Lung Cancer Centre, Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoffer LJ, Robitaille L, Swinton N, Agulnik J, Cohen V, Small D, Pepe C, Eintracht S. Appropriate vitamin D loading regimen for patients with advanced lung cancer. Nutr J. 2016 Oct 6;15(1):84. doi: 10.1186/s12937-016-0203-8. PMID 27716304